CLINICAL TRIAL: NCT00651053
Title: Validation of Endoscopic Ultrasound Criteria for Diagnosis of Chronic Pancreatitis Using Dual Secretin and Cholecystokinin Pancreatic Function Testing as Reference Standard
Brief Title: Endoscopic Ultrasound Compared With Pancreatic Function Testing for Diagnosis of Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: ChiRhoClin, Inc. (Industry); The National Pancreas Foundation (Other)
Responsible Party: Tyler Stevens, M.D., Cleveland Clinic Foundatino
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: CRC 2005-01
Record Dates: First submitted 2008-03-30; First posted 2008-04-02 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2008-03

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EUS — Sensitivity and specificity of EUS will be compared with PFT as reference standard.

SUMMARY:
This is a investigator-initiated, single-center, prospective study to evaluate endoscopic ultrasound (EUS) as a diagnostic test for chronic pancreatitis (CP). EUS detects abnormalities of the pancreas that may represent scarring from CP. The validation of any new test requires a comparison with the best available reference standards. There is no true "gold standard" for diagnosis of CP; however, pancreatic function testing (PFT) is highly sensitive for exocrine dysfunction as a surrogate for early fibrosis, and is widely considered the non-histologic gold standard. There are no well-designed prospective studies comparing EUS with PFT as reference standard.

EUS detects parenchymal and ductal features of CP said to correlate with fibrosis. We hypothesize that a predominance of parenchymal fibrosis results in diminished acinar-cell secretion of enzymes. Conversely, a predominance of ductal fibrosis results in impairment of ductal secretion of bicarbonate. Because secretin and cholecystokinin (CCK) PFTs measure unique aspects of pancreatic function (duct-cell and acinar-cell function, respectively), the use of both hormonal stimulants will allow the most comprehensive investigation of the significance of EUS features. There are no studies comparing EUS with combined or dual performance of secretin and CCK PFTs.

The primary objective of this study is to determine the test characteristics of EUS for diagnosis of CP compared with dual secretin- and CCK- stimulated PFTs as reference standard. Secondary objectives include to: 1. Determine the optimal number and relative functional importance of specific EUS criteria, 2. Compare the test characteristics of linear- and radial-array EUS.

190 patients evaluated for pancreatitis or pancreatic-type abdominal pain will undergo the "new test" (radial and linear EUS) and the reference standard (CCK and secretin PFTs). The EUS examinations will be videotaped and interpreted in a blinded fashion. EUS scores will be compared with PFT results to allow the calculation of sensitivity and specificity of linear and radial EUS. Receiver operating characteristics (ROC) analysis will be used to determine the optimal number of EUS criteria for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age greater than 18 years.
2. Capable of informed consent.
3. If female and not more than 1 year post-menopausal, or surgically sterile, must use medically accepted form of contraception or abstain from sexual activities during study.
4. EUS and CCK ePFT planned for a structural evaluation of the pancreas in patients with pancreatitis or pancreatic-type abdominal pain.

Exclusion Criteria:

1. Severe cardiac disease (stable or unstable angina, congestive heart failure, uncontrolled arrhythmias, implantable defibrillator, severe valvular disease, etc.).
2. Severe pulmonary disease (Severe asthma, COPD or interstitial lung disease requiring nebulizer treatment or home oxygen, pulmonary hypertension).
3. Severe renal disease (history of chronic renal insufficiency [creatinine >2.0] or chronic hemodialysis).
4. Inability to undergo conscious sedation or general anesthesia.
5. Ongoing illicit drug use or abuse. Must be drug free for >1 year.
6. Acute pancreatitis within the past 2 months.
7. Prior pancreatic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-05; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of EUS

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States